CLINICAL TRIAL: NCT03659942
Title: Study of the Cannabis Use of Minors Imprisoned in the PACA Region (France)
Brief Title: Study of the Cannabis Use of Minors Imprisoned in the PACA Region
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-25
Record Dates: First submitted 2018-09-04; First posted 2018-09-06 (Actual); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Cannabis Use

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experimental group: New child arriving in detention CAST questionnaire will be performed
  Interventions: Other: CAST questionnaire

INTERVENTIONS:
Other: CAST questionnaire — the CAST questionnaire will be used to answer the main objective of the study and to identify consumers with problematic cannabis use. This is a validated self-questionnaire in France (Legleye et al., 2011), specific to the adolescent population, which is interpreted according to the score obtained (Bastiani et al., 2013, Legleye et al. 2007, Legleye et al., 2011). It includes 6 items with answer modes coded from 0 to 4. The total score obtained by summing these 6 items can therefore vary from 0 to 24. We define users without risk for a score of less than 3, users with low risk for a score greater than or equal to 3 and less than 7, and finally those with a risk of problematic use for a score greater than or equal to 7

SUMMARY:
To date, there is little data on the consumption of young adults in detention.

The main objective of this project is to document the prevalence of problematic cannabis use before incarceration among juveniles detained in the various detention centers in the PACA

Secondary objectives are to document:

* the prevalence of cannabis use over the course of life, last year and last month;
* the prevalence of harm and risky behavior associated with the use of a psychoactive substance
* associated addictions and first and foremost tobacco
* the determinants (socio-demographic, socio-economic, environmental, etc.) of problem use and cannabis use.

This is a multicenter cross-sectional study aimed at establishing an exhaustive picture of the defined population region over a 12-month period.

The holder of the parental authority exercise and the individual agreeing to participate in the study must:

* sign an informed consent a no objection card
* complete a car book and hetero-questionnaires. The time of handover is evaluated at 30 minutes.

The CAST questionnaire will be used to answer the main purpose of the study and to identify consumers with problematic cannabis use.

CAST scores will be calculated. Abnormal CAST proportions will be presented along with their 95% confidence intervals. The links between the score and the various variables identified as determinants will be tested using uni and multivariate analyzes.

The assessment of the health status and needs of this extremely vulnerable population is a prerequisite for defining specific regional objectives and for establishing a coherent and coordinated effective health intervention within the community. prisoner in France.

DETAILED DESCRIPTION:
To date, there is little data on the consumption of young adults in detention when they are the first consumers in the general population in France and they represent a particularly vulnerable population within the prison population.

objectives The main objective of this project is to document the prevalence of problematic cannabis use before incarceration among juveniles detained in the various detention centers in the P.A.C.A.

Secondary objectives are to document:

* the prevalence of cannabis use over the course of life, last year and last month;
* the prevalence of harm and risky behavior associated with the use of a psychoactive substance
* associated addictions and first and foremost tobacco
* the determinants (socio-demographic, socio-economic, environmental, etc.) of problem use and cannabis use.

Method This is a multicenter cross-sectional study aimed at establishing an exhaustive picture of the defined population (juvenile detainees in the P.A.C.A.) region over a 12-month period.

The holder of the parental authority exercise and the individual agreeing to participate in the study must:

* sign an informed consent a no objection card
* complete a car book and hetero-questionnaires. The time of handover is evaluated at 30 minutes.

The CAST questionnaire will be used to answer the main purpose of the study and to identify consumers with problematic cannabis use.

CAST scores will be calculated. Abnormal CAST proportions will be presented along with their 95% confidence intervals. The links between the score and the various variables identified as determinants (socio-demographic, socio-economic, environmental, other addictions, etc.) will be tested using uni and multivariate analyzes.

Expected results The assessment of the health status and needs of this extremely vulnerable population is a prerequisite for defining specific regional objectives and for establishing a coherent and coordinated effective health intervention within the community. prisoner in France.

ELIGIBILITY:
Inclusion Criteria:

* Newcomer subject in detention,
* Subject having been informed about the study and not expressing opposition to participating in the study.
* Legal officer who was informed about the study and did not express any opposition to participate in the study.
* Subject including French and able to fill self-questionnaires, and not presenting attacks of the severe cognitive functions

Exclusion Criteria:

Subject already incarcerated less than 6 months before its inclusion,

* subject with severe hearing loss,
* Subject not having agreed to participate in the study,
* Holder of parental authority who has not given his consent,
* Subject not including French.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients new arriving in prison
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-01 (Estimated); Primary Completion 2020-01 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
CAST questionnaire score | 30 minutes
  the CAST questionnaire will be used to answer the main objective of the study and to identify consumers with problematic cannabis use. This is a validated self-questionnaire in France (Legleye et al., 2011), specific to the adolescent population, which is interpreted according to the score obtained. It includes 6 items with answer modes coded from 0 to 4. The total score obtained by summing these 6 items can therefore vary from 0 to 24. We define users without risk for a score of less than 3, users with low risk for a score greater than or equal to 3 and less than 7, and finally those with a risk of problematic use for a score greater than or equal to 7

CONTACTS AND LOCATIONS:
Overall Officials: EMILIE GARRIDO PRADALIE, Study Director — APHM
Locations (1):
- Assistance Publique Des Hopitaux de Marseille, Marseille, PACA, France